CLINICAL TRIAL: NCT06525792
Title: A Clinical Study on Ozone Autohemotherapy for the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Heyun Cheng, Study Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHGJ20190414
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Cerebrovascular Disease
MeSH Terms: interventions — Oxygen; Ozone; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Standard treatment
  Interventions: Procedure: Standard therapy
- Experimental group 1 (Experimental)
  Interventions: Procedure: Oxygen
- Experimental group 2 (Experimental)
  Interventions: Procedure: Ozone

INTERVENTIONS:
Procedure: Oxygen — Oxygen and standard therapy were given
  Arms: Experimental group 1
Procedure: Ozone — Ozone and standard therapy were given
  Arms: Experimental group 2
Procedure: Standard therapy — Best standard of care
  Arms: Control group

SUMMARY:
Clinical studies applying ozonated autohemotherapy to treat acute cerebrovascular diseases have validated the safety and efficacy of this treatment, as well as explored its mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by cranial CT or MRI examination, first-ever stroke, hospital admission within <24 hours of symptom onset,
2. age >18 years,
3. NIHSS score between 4 and 15,
4. TOAST classification as large artery atherosclerosis,
5. complete clinical records, minimum follow-up period of ≥3 months post-discharge,
6. willingness to undergo brachial blood puncture treatment, and provision of informed consent

Exclusion Criteria:

1. other neurological disorders, cerebral infarction caused by vertebral-basilar artery disease, cardioembolic stroke, or large-vessel vasculitis, acute or chronic infectious diseases, autoimmune or hematologic disorders, malignant tumors, mental abnormalities, severe heart, liver, or kidney dysfunction, intracerebral hemorrhage, and craniocerebral surgery history.
2. Contraindications for ozone therapy included hyperthyroidism, favism, severe coagulation disorders, and abnormal puncture site barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The expression of SOD(Superoxide dismutase) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China